CLINICAL TRIAL: NCT00942422
Title: The Clinical and Biologic Evaluation of Polyphenon E, an Extract of Green Tea Containing EGCG, in Plasma Cell Dyscrasias - Pilot Study
Brief Title: Green Tea Extract in Treating Patients With Monoclonal Gammopathy of Undetermined Significance and/or Smoldering Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual and early termination
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Zonder, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000646899; P30CA022453 (NIH); WSU-2009-015 (Other: Barbara Ann Karmanos Cancer Institute); NCT01589887 (obsolete NCT alias)
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm; Precancerous Condition
Keywords: monoclonal gammopathy of undetermined significance; smoldering multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma | interventions — Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- defined green tea catechin extract / correlative analysis (Experimental): Polyphenon E, an oral capsule form of EGCG extracted from green tea, 800 mg administered daily on an empty stomach (at least 1 hour before or 2 hrs after a meal)Patients receive oral green tea catechin extract (Polyphenon E) daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: defined green tea catechin extract; Genetic: gene expression analysis; Genetic: protein analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Dietary Supplement: defined green tea catechin extract — Polyphenon E, an oral capsule form of EGCG extracted from green tea, 800 mg administered daily on an empty stomach (at least 1 hour before or 2 hrs after a meal)Patients receive oral green tea catechin extract (Polyphenon E) daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Genetic: gene expression analysis — Blood and bone marrow samples will be obtained prior to the start of treatment and at the conclusion of the study for correlative studies. An additional peripheral blood sample will be obtained on day 8 of the first cycle of therapy.
Genetic: protein analysis — Blood and bone marrow samples will be obtained prior to the start of treatment and at the conclusion of the study for correlative studies. An additional peripheral blood sample will be obtained on day 8 of the first cycle of therapy.
Other: laboratory biomarker analysis — Blood and bone marrow samples will be obtained prior to the start of treatment and at the conclusion of the study for correlative studies. An additional peripheral blood sample will be obtained on day 8 of the first cycle of therapy.

SUMMARY:
RATIONALE: Green tea extract contains ingredients that may prevent or slow the growth of monoclonal gammopathy of undetermined significance and/or smoldering multiple myeloma.

PURPOSE: This phase II trial is studying how well green tea extract works in treating patients with monoclonal gammopathy of undetermined significance and/or smoldering multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Conduct a pilot study investigating the effects of Polyphenon E, a compound extracted from green tea which contains epigallocatechin-3-gallate (EGCG), on monoclonal protein levels in patients with monoclonal gammopathy of undetermined significance and/or smoldering multiple myeloma.

Secondary

* Collect, process, and store blood and marrow specimens for future measurement of the biologic effects of Polyphenon E on the plasma cells of these patients by utilizing proteosome activity assays and gene expression profiling.

OUTLINE: Patients receive oral green tea catechin extract (Polyphenon E) daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients may undergo blood, urine, and bone marrow sample collection periodically for correlative laboratory studies. Samples are analyzed for monoclonal protein (M-protein) levels, proteosome function, and gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Measurable monoclonal protein in the serum (for immunoglobin [Ig]G or IgM, >= 1.0 g/dL using serum protein electrophoresis [SPEP]/immunofixation electrophoresis [IFE]; for IgA, an SPEP/IFE confirming the presence of a monoclonal IgA band plus a quantitative IgA level of >= 750 mg/dL) OR measurable urine Bence Jones paraprotein (>= 500mg/24hrs) OR a measurable serum free light chain (FLC), defined as an involved FLC level of >10 mg/dl, and a serum FLC ratio that is abnormal
* Neutrophil count >= 1,500
* Platelet count >= 100,000
* Hemoglobin >= 9mg/dL
* Alanine aminotransferase (ALT) =< institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) =< IULN
* Total bilirubin =< IULN
* Alkaline phosphatase =< IULN
* Any ethnic group
* Prior therapy is allowed if >= 4 weeks prior to registration
* Life expectancy of at least 6 months
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to comply with oral home treatment and visit schedule
* Patients with reproductive capacity must be willing to use adequate contraception (barrier contraception, birth control pills, or other highly effective hormonal agents) or abstain from sexual activity for the duration of the study and 30 days beyond the end of therapy

Exclusion Criteria:

* Pregnant women
* Breastfeeding women
* Confirmed symptomatic multiple myeloma (MM), defined by any of the following:
* Lytic lesions on skeletal survey
* Anemia attributable to plasma cell infiltrate in marrow
* Hypercalcemia
* Renal dysfunction not attributable to other causes
* Uncontrolled intercurrent illness, including but not limited to active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness or social situations that would compromise compliance with study medication or follow up visits
* Patients with high predisposition to gastrointestinal bleeding, such as known gastroesophageal varices or active peptic ulcer disease
* Patients with chronic liver disease (such as hepatitis B, hepatitis C, or alcoholic cirrhosis)
* Prior daily ingestion of green tea or green tea extract within 6 months of study entry
* Patients who have previously experienced any adverse symptoms related to green tea or any of the inactive components present in Polyphenon E capsules
* Concurrent use of investigational or commercial agent or therapy with the intent to treat MGUS and/or SMM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Zonder, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Defined Green Tea Catechin Extract / Correlative Analysis
Started | 8
Completed | 5
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Progressive diease | 1

BASELINE CHARACTERISTICS:
Groups:
- Defined Green Tea Catechin Extract / Correlative Analysis: Polyphenon E, an oral capsule form of EGCG extracted from green tea, 800 mg administered daily on an empty stomach (at least 1 hour before or 2 hrs after a meal). Patients receive oral green tea catechin extract (Polyphenon E) daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Defined Green Tea Catechin Extract / Correlative Analysis
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Sustained M-protein Reduction of ≥ 25% From Baseline
Description: This is a monthly blood test, done at the beginning of each cycle of therapy. The M-protein is a surrogate marker routinely used to estimate the degree of plasma cell cyto-reduction brought about by therapy. In active multiple myeloma, a 25% reduction in the M-protein level would correspond to a "minor response," an improvement recognized as having some clinical benefit.
Time Frame: Day one of each 28-day cycle for a total of up to 6 cycles
Measure: Number; unit: percentage of patients
Groups:
- Defined Green Tea Catechin Extract / Correlative Analysis: Polyphenon E, an oral capsule form of EGCG extracted from green tea, 800 mg administered daily on an empty stomach (at least 1 hour before or 2 hrs after a meal)Patients receive oral green tea catechin extract (Polyphenon E) daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  defined green tea catechin extract: Polyphenon E, an oral capsule form of EGCG extracted from green tea, 800 mg administered daily on an empty stomach (at least 1 hour before or 2 hrs after a meal)Patients receive oral green tea catechin extract (Polyphenon E) daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  gene expression analysis: Blood and bone marrow samples will be obtained prior to the start of treatment and at the conclusion of the study for correlative studies. An additional peripheral blood sample will be obtained on day 8 of the
Arm/Group | Defined Green Tea Catechin Extract / Correlative Analysis
Number analyzed (Participants) | 8
percentage of patients | 0

ADVERSE EVENTS:
Groups:
- Defined Green Tea Catechin Extract / Correlative Analysis: Polyphenon E, an oral capsule form of EGCG extracted from green tea, 800 mg administered daily on an empty stomach (at least 1 hour before or 2 hrs after a meal)Patients receive oral green tea catechin extract (Polyphenon E) daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  gene expression analysis: Blood and bone marrow samples will be obtained prior to the start of treatment and at the conclusion of the study for correlative studies. An additional peripheral blood sample will be obtained on day 8 of the
Arm/Group | Defined Green Tea Catechin Extract / Correlative Analysis
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Defined Green Tea Catechin Extract / Correlative Analysis (N=8)
Hyperglycemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Defined Green Tea Catechin Extract / Correlative Analysis (N=8)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Reflux (Gastrointestinal disorders) | 1 (1)
Loose Stools (Gastrointestinal disorders) | 3 (3)
Difficulty Swallowing Pills (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Increased ALT (Metabolism and nutrition disorders) | 2 (2)
Increased AST (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (4)
Increased Creatinine (Metabolism and nutrition disorders) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Palpable left axillary and mandibular lymph nodes (Skin and subcutaneous tissue disorders) | 1 (1)
Brusing left arm (Skin and subcutaneous tissue disorders) | 1 (1)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1)
Jock Itch (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Viral Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post Nasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Heart Palpitation (Cardiac disorders) | 1 (1)
Borderline bradycardia (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Insomnia (General disorders) | 1 (1)
Night sweats (General disorders) | 1 (1)
Weight Gain (General disorders) | 1 (1)
Belching (General disorders) | 1 (1)
Skin Redness (General disorders) | 1 (1)
Mood Changes (Nervous system disorders) | 1 (1)
Ankle Tenderness/Pain (General disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Back Pain (General disorders) | 2 (2)
Chest Pain (General disorders) | 1 (1)
Cramping in neck (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Low accrual and early termination limits the conclusions one could draw. Although no pts on this trial met the primary endpoint of a 25% or greater M-protein reduction, the small number of pts enrolled prohibits formal statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No